CLINICAL TRIAL: NCT02064283
Title: Early Assessment of Treatment Response Using Functional Diffusion Mapping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: UMCC 2006.111; HUM00009498 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2014-02-13; First posted 2014-02-17 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diffusion MRI Assessment (Experimental): Men with newly diagnosed metastatic disease initiating therapy with androgen deprivation, or men with hormone refractory prostate cancer initiating treatment with chemotherapy, will be assessed by diffusion MRI (Magnetic Resonance Imaging) at baseline, 2 weeks and again at 9-12 weeks.
  Interventions: Procedure: Diffusion MRI

INTERVENTIONS:
Procedure: Diffusion MRI

SUMMARY:
This study will evaluate the feasibility of identifying changes in diffusion MRI characteristics of bone that correlates with response to therapy in men with metastatic prostate cancer.

DETAILED DESCRIPTION:
This study will evaluate a special type of MRI (magnetic resonance imaging) scan that measures the movement of water molecules through tissue called diffusion MRI. Researchers are using this new MRI technology to track the diffusion, or movement, of water through tumor tissue, and map these changes as a cancer patient undergoes treatment. Early research seems to indicate that tumor cells restrict the movement of water, so as tumor cells die, the movement of water changes within the tumor. These changes in the movement (diffusion) of water may help doctors determine earlier than traditional tests whether a patient's cancer is responding (getting better) to treatment. This study will evaluate the feasibility of identifying changes in diffusion MRI characteristics of bone that correlates with response to therapy in men with metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of prostate cancer.
* Evidence of metastatic disease by bone scan.
* Patients must be initiating systemic therapy for metastatic disease.
* New D2 disease beginning therapy with androgen deprivation.
* CRPC (Castration Resistant Prostate Cancer) beginning systemic non hormonal therapy.
* Patients must be willing to provide the blood samples for the correlative markers.
* Patients must be able to lie flat in an MRI (Magnetic Resonance Imaging) magnet for 30-60 minutes.
* Life expectancy of 12 weeks or greater.
* All patients must be informed of the investigational nature of this study and must sign an informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Contraindication to MRI imaging.
* Patients who require sedation with general anesthesia to undergo MRI imaging.
* Weight greater than 275 pounds.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change in diffusion MRI measurements | Baseline, 2 weeks and 9-12 weeks
  Identify changes in Diffusion Magnetic Resonance Imaging (MRI) measurements and correlate the changes with response to therapy.

SECONDARY OUTCOMES:
Change in units/L of CK18Asp306 | Baseline, 2 weeks and 9-12 weeks
  Levels of CK18Asp396 can be measured in serum using a commercially available ELISA (Enzyme-linked Immunosorbent Assay). Changes in serum CK18Asp396 (a marker of apoptosis) will be correlated with functional diffusion maps and treatment response.
Change in levels of bone turnover markers | Baseline, 2 weeks and 9-12 weeks
  Correlate the changes in biochemical markers of bone turnover, such as N-telopeptide and bone-specific alkaline phosphatase, with functional diffusion maps and treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Maha Hussain, MD, FACP, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Brisset JC, Hoff BA, Chenevert TL, Jacobson JA, Boes JL, Galban S, Rehemtulla A, Johnson TD, Pienta KJ, Galban CJ, Meyer CR, Schakel T, Nicolay K, Alva AS, Hussain M, Ross BD. Integrated multimodal imaging of dynamic bone-tumor alterations associated with metastatic prostate cancer. PLoS One. 2015 Apr 10;10(4):e0123877. doi: 10.1371/journal.pone.0123877. eCollection 2015. PMID 25859981